CLINICAL TRIAL: NCT05026801
Title: A Randomized, Double-blinded Phase 3 Multi-center Study of the Clinical and Microbiologic Efficacy of a Combination of Azithromycin and Hydroxychloroquine for Treatment of COVID-19 Infection
Brief Title: Azithromycin Plus Hydroxychloroquine for COVID-19 Infection
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Inadequate support to carry out study
Sponsor: Iterum Therapeutics, International Limited (Industry)
Collaborators: Waterbury Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IT005-501
Record Dates: First submitted 2021-02-08; First posted 2021-08-30 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Respiratory Tract Infection Viral
Keywords: Coronavirus
MeSH Terms: conditions — Coronavirus Infections | interventions — Azithromycin; Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Approximately 200 patients with symptoms of a RTI who test positive for SARS-CoV-2 by polymerase chain reaction (PCR) will receive a combination of azithromycin 500 mg and chloroquine 500 mg or matching placebos for six consecutive days. There will be two treatment regimens into which patients are randomized so that all patients will receive some active therapy. A sequential probability ratio test will be employed in which comparisons between each regimen will be made with every Day 3 PCR endpoint; if the p value crosses a p=0.001 threshold for any pairwise comparison, the less efficacious arm will be closed to further enrollment and superiority will be declared.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Azithromycin plus hydroxychloroquine (Active Comparator): Azithromycin 500 mg plus hydroxychloroquine 600 mg by mouth daily for six consecutive days
  Interventions: Drug: Azithromycin plus hydroxychloroquine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Azithromycin plus hydroxychloroquine

INTERVENTIONS:
Drug: Azithromycin plus hydroxychloroquine — All patients will receive active comparator. One group will receive placebo on D1-3 followed by active comparator D4-9, while the other group will receive active comparator D1-6 followed by placebo D7-9.
  Other Names: Placebo

SUMMARY:
This is a randomized, double-blinded, Phase 3, multi-center trial of the clinical and microbiologic response of patients with a respiratory tract infection (RTI) due to coronavirus treated with a combination of azithromycin and hydroxychloroquine.

Approximately 200 patients with symptoms of an RTI who test positive for SARS-CoV-2 by polymerase chain reaction (PCR) will receive a combination of azithromycin 500 mg and hydroxychloroquine 600 mg or matching placebos for six consecutive days. There will be two treatment regimens into which patients are randomized so that all patients will receive some active therapy.

DETAILED DESCRIPTION:
As of March 22, 2020, a total of 311,988 people worldwide have been diagnosed with a respiratory infection caused by SARS-CoV-2 of whom 13,407 have died. In the United States 26,747 patients have tested positive of whom 340 have died. There is at present no established therapy for this infection. After the SARS epidemic in 2002, investigations identified chloroquine as a possible inhibitor of replication of this coronavirus. When the SARS-CoV-2 epidemic started in December of 2019, clinicians began to use chloroquine in an attempt to control the infection in newly diagnosed patients. Investigators from China reported chloroquine phosphate has apparent efficacy in treatment of pneumonia due to SARS-CoV-2. Following this report, investigators in France initiated an open label study of hydroxychloroquine, with the addition of azithromycin, in a small number of subjects with SARS-CoV-2 infection. Relative to no treatment the investigators identified a significant reduction in viral isolation by PCR in the nasal swabs of treated patients, with an additional effect seen when patients were also given azithromycin. Azithromycin, like chloroquine, is a weak base that concentrates in endosomes and lysosomes and raises the pH in those vesicles. It is possible that azithromycin and chloroquine's effect on endosomal processing reduces the inflammatory response by affecting TLR4 signaling through the endosomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years of age
2. History of a respiratory tract infection (RTI) for more than one but less than six days including two or more of the following signs and symptoms of an RTI:

   • Fever (T ≥ 38.0 C, 100.5 F), cough, sputum production, arthralgia/myalgia, anosmia/ageusia or difficulty breathing.
3. A nasal or throat swab or nasal wash positive by PCR for SARS-CoV-2.
4. Has given written informed consent to participate in the study. Due to the public health issues related to this viral infection, witnessed informed consent may be obtained remotely.

Exclusion Criteria:

Exclusion Criteria:

1. Patients likely, in the opinion of the investigator, to require hospitalization within 48 hours of randomization into the study.
2. Concurrent use of non-study antibacterial drug therapy that would have a potential effect on outcome evaluations in patients with an RTI
3. Concurrent use of any other medications for the purpose of treating a viral infection such as influenza antivirals
4. Inability to swallow oral medication in tablet form
5. Patient has severe chronic kidney disease, or is receiving hemodialysis, or peritoneal dialysis or had a renal transplant
6. Patient is known to have severe neutropenia
7. Patients with a known prolongation of the QT interval or are taking medications which could prolong the QT interval
8. Patient is known to be pregnant
9. Patients with a known history of myasthenia gravis
10. Patients with a history of allergy to azithromycin, hydroxychloroquine or chloroquine
11. Patient is considered unlikely to survive the study period or has a rapidly progressive or terminal illness, including septic shock, associated with a high risk of mortality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2021-08-26 (Actual)

PRIMARY OUTCOMES:
Microbiologic response | Day 3 (+/- 1 day)
  Presence or absence of SARS-CoV-2 by PCR on nasopharyngeal specimen

SECONDARY OUTCOMES:
Combined clinical and microbiologic response | Day 3 (+/- 1 day)
  Presence or absence of SARS-CoV-2 by PCR on nasopharyngeal specimen and improvement in at least two of the signs and symptoms of RTI

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dunne, MD, Principal Investigator — Iterum Therapeutics
Locations (1):
- Waterbury Hospial, Waterbury, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 30 days of study completion.
Access Criteria: Data access requests will be reviewed on a case by case basis. Requestors will be required to sign a Data Access Agreement.
URL: http://www.iterumtx.com